CLINICAL TRIAL: NCT03181321
Title: The First Twenty for Volunteer Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Development and Research Institutes, Inc. (Other)
Responsible Party: Principal Investigator, Rena Sue Day, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-14-0749; EMW-2013-FP-00983 (Other: FEMA)
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Obesity; Cardiovascular Diseases; Occupational Injuries
Keywords: nutrition; fitness; cardiovascular disease; firefighters; obesity; injury
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Occupational Injuries; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a 6 month, two-arm, CRCT: TF20 vs. Control (which will receive delayed treatment after 6 months). Eligible fire departments volunteering for the trial will be randomized to one of the two study treatment arms. Treatment outcomes will be assessed at baseline and 6 months by our staff.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The First Twenty (Experimental): The TF20 incorporates individual goal setting and health coaching, leveraging cultural aspects of the fire service and group cohesion to motivate behavior change. The TF20 focuses on the unique needs of FF with culturally relevant nutrition and fitness strategies. TF20 was primarily designed as a cost-effective, stand-alone program for departments which have no health promotion initiative. Program components include practical approaches to nutrition, fitness and mental health.
  Interventions: Behavioral: The First Twenty
- Control (No Intervention): Participants in this arm will not be asked to change anything in their lifestyle during the 6 month period.

INTERVENTIONS:
Behavioral: The First Twenty — The TF20 incorporates individual goal setting and health coaching, leveraging cultural aspects of the fire service and group cohesion to motivate behavior change. The TF20 focuses on the unique needs of FF with culturally relevant nutrition and fitness strategies. TF20 was primarily designed as a cost-effective, stand-alone program for departments which have no health promotion initiative. Program components include practical approaches to nutrition, fitness and mental health.
  Arms: The First Twenty

SUMMARY:
The purpose of this study is to assess the efficacy of an internet-based firefighter health and wellness program for volunteer fire departments.

DETAILED DESCRIPTION:
A national sample of volunteer fire departments will be recruited for a 6 month, CRCT with a cross-over treatment design to determine the efficacy of The First Twenty (TF20), a wellness program focused on nutrition and fitness for firefighters. Modifications to the existing TF20 will be made to enhance the health coaching features and include tools for program evaluation. Study outcomes (changes in weight, BMI, body fat percentage, waist circumference, dietary intakes, blood pressure, and fitness activities) will be assessed pre- and post-intervention.

This will be the first internet-based, occupationally tailored health and wellness program implemented for the volunteer fire service. TF20 will be an essential cost effective tool to address the epidemic of unhealthy body composition, nutrition and fitness among firefighters.

ELIGIBILITY:
Inclusion Criteria:

* first responder within a participating fire department
* willing to complete all assessments
* internet accessibility through a computer, tablet or smartphone and ability to use devices appropriately

Exclusion Criteria:

- not a first responder within a participating fire department

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | baseline, 6 months
  BMI from measured height and weight
Change in Body Fat Percentage | baseline, 6 months
  body fat % from Tanita scale measurement
Change in Waist Circumference | baseline, 6 months
  waist circumference from measured waist using a tape

SECONDARY OUTCOMES:
Change in Food and nutrient intake as assessed by the Food Frequency Questionnaire (FFQ) | baseline, 6 months
  The Food and Frequency Questionnaire (FFQ) is a self-administered, semi-quantitative, food frequency questionnaire developed by the principal investigator. The FFQ presents a food list, which contains items contributing most to selected nutrient intakes among firefighters and foods encouraged by the intervention. FFQ data will be used to calculate usual nutrient intakes using the Food Intake Analysis System (FIASMe).
Change in self reported physical activity and inactivity | baseline, 6 months
  SRPA

CONTACTS AND LOCATIONS:
Overall Officials: Rena S Day, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No